CLINICAL TRIAL: NCT03695900
Title: Impact of Arterial Oxygen Saturation Range on Ventilatory Stability in Extremely Premature Infants
Brief Title: Arterial Oxygen Saturation on Ventilatory Stability in Extremely Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Gerber Foundation (Other)
Responsible Party: Principal Investigator, Nelson Claure, Associate Professor of Pediatrics, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20180536
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Apnea of Prematurity; Desaturation of Blood; Central Apnea; Periodic Breathing; Obstructive Apnea of Newborn
MeSH Terms: conditions — Apnea; Sleep Apnea, Central

STUDY DESIGN:
Intervention Model Description: This is a prospective crossover study to compare the within-subject effect of the two target ranges of arterial oxygen saturation (SpO2, 93-95% vs 90-92%) on ventilatory stability in premature infants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeting SpO2 at 93-95% followed by targeting at 90-92% (Other): FiO2 adjusted to keep basal SpO2 at target range of 93-95% for 2 hours, followed by FiO2 adjusted to keep basal SpO2 at target range of 90-92% for 2 hours.
  Interventions: Other: Targeting SpO2 at 93-95%; Other: Targeting SpO2 at 90-92%
- Targeting SpO2 at 90-92% followed by targeting at 93-95% (Other): FiO2 adjusted to keep basal SpO2 at target range of 90-92% for 2 hours, followed by FiO2 adjusted to keep basal SpO2 at target range of 93-95% for 2 hours.
  Interventions: Other: Targeting SpO2 at 93-95%; Other: Targeting SpO2 at 90-92%

INTERVENTIONS:
Other: Targeting SpO2 at 93-95% — FiO2 adjusted to keep basal SpO2 at target range of 93-95% for 2 hours
Other: Targeting SpO2 at 90-92% — FiO2 adjusted to keep basal SpO2 at target range of 90-92% for 2 hours.

SUMMARY:
This is a prospective crossover study to compare the within-subject effect of the two target ranges of arterial oxygen saturation (SpO2), both within the clinically recommended range of 90- 95%. The specific objective of this study to evaluate the impact of targeting SpO2 within 93-95% compared to the 90-92% range on ventilatory stability in premature infants of 23-29 weeks gestational age (GA).

ELIGIBILITY:
Inclusion Criteria:

* 23 0/7- 29 6/7 weeks gestational age
* Postnatal age ≥ 14 days
* Requiring FiO2 ≥ 0.25 to keep SpO2 90-95%
* Parental informed consent

Exclusion Criteria:

* Severe congenital anomalies that may affect pulmonary or neurosensory development
* Severe CNS pathology that may alter respiratory control function

Max Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
ventilatory stability by frequency of central apnea | 2 hours
  by frequency of central apnea
ventilatory stability by frequency of obstructive apnea | 2 hours
  by frequency of obstructive apnea
ventilatory stability by density of periodic breathing | 2 hours
  by density of periodic breathing
ventilatory stability by time series of inter-breath intervals | 2 hours
  by time series of inter-breath intervals

SECONDARY OUTCOMES:
oxygenation stability by frequency of intermittent hypoxemia episodes | 2 hours
  frequency of episodes with SpO2 < 80%
frequency of bradycardia episodes | 2 hours
  frequency of episodes with HR < 100 bpm

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Claure, MSc, PhD, Principal Investigator — University of Miami; Eduardo Bancalari, MD, Principal Investigator — University of Miami; Deepak Jain, MD, Principal Investigator — University of Miami; Waleed Kurtom, MD, Principal Investigator — Jackson Health System
Locations (1):
- Holtz Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurtom W, Dormishian A, Jain D, Schott A, Aguilar AC, Grieb G, Bancalari E, Claure N. Effect of the Target Range on Arterial Oxygen Saturation Stability in Extremely Premature Infants. Neonatology. 2022;119(5):638-643. doi: 10.1159/000525271. Epub 2022 Aug 26. PMID 36030769